CLINICAL TRIAL: NCT05573542
Title: Early Signs of Parkinson's Disease Pathology in the Colon of Patients With Irritable Bowel Syndrome
Brief Title: Early Signs of Parkinsons Disease in IBS
Status: Enrolling by invitation | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: VHIR (Unknown); Aston University (Other); Region Örebro County (Other)
Responsible Party: Principal Investigator, Robert Brummer, Professor, MD, Örebro University, Sweden
Other Study IDs: PARKIBS
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease; Irritable Bowel Syndrome
Keywords: Alpha-synuclein; Intestinal permeability; Gut-brain axis; Mucosal ultrastructure; Brain function; Microbiota; Metabolomics
MeSH Terms: conditions — Parkinson Disease; Irritable Bowel Syndrome; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Parkinson's: Individuals with confirmed diagnosis of Parkinson's disease by neurologist.
- Patients with irritable bowel syndrome: Individuals with IBS according to ROME IV criterias
- Healthy controls: Healthy individuals lacking both IBS and Parkinson's disease, in addition to other criteras stated in the Eligibility section.

SUMMARY:
Bowel symptoms like constipation and abdominal pain are characteristic symptoms of irritable bowel syndrome (IBS). The pathogenesis and pathophysiology are not fully understood but subject to intense research, with emphasis on aberrations in the gut-brain axis, low-grade inflammation and gut barrier dysfunction that results in increased permeability and microbial translocation. Many patients with Parkinson's disease (PD) have reported bowel symptoms similar to that in IBS patients decades prior to the diagnosis of PD. Epidemiological studies show a significantly elevated risk of developing PD in IBS patients, though there is no knowledge on a pathogenic connection between these disorders. Recent studies show increased gut permeability and intestinal presence of pathological alpha-synuclein aggregates, the neuropathological hallmark in PD, indicating the involvement of the gut-brain axis. We aim to compare the presence of colonic alpha-synuclein between IBS, PD patients and healthy controls to relate these findings to intestinal permeability, ultrastructural mucosal changes, immune cell interactions, microbiota composition and brain function. This project could identify IBS groups at risk of developing PD and birth the development of early clinical diagnostic methods.

DETAILED DESCRIPTION:
All study participants will give 3 study visits and questionnaires and faecal collection kits will be sent to them before the first visit.

Visit 1: Study participants will undergo a sigmoidoscopy during which the researchers will collect 16 biopies. Twelve of the biopsies goes to ussing chamber studies of permeability while the remaining biopsies will be alliqoted for ultrastructural characterisation, alpha-synuclein aggregation assay and immunoflourescence. Blood samples will be drawn from the participants at this visits for metabolomic studies and platelet aggregation potential. In addition, study participants will also bring filled out questionnaires and faecal samples (microbiota analysis).

Visit 2: Study participants will undergo a functional magnetic resonance imaging session for analysis of brain function. This visit will last for approximately 1 hour (preparations included).

Visit 3: Participants will come in for a final sigmoidoscopy where the biopsies will be collected exclusively for performing the immuno-neurophenotyping of lamina propria lymphocytes.

ELIGIBILITY:
Patients with Parkinson's disease

Inclusion Criteria:

1. Confirmed diagnosis by neurologist
2. Males or females aged 45-85 years
3. Signed informed consent

Exclusion Criteria:

1. Other confirmed GI diseases (such as inflammatory bowel diseases)
2. Concurrent or recent treatment with antibiotics (< 12 weeks)
3. Concurrent or recent (< 4 weeks) use of nutritional supplements or herb products affecting intestinal function or mood (e.g. aloe vera, St. John´s Wort and probiotics/prebiotics).
4. Diagnosis of major psychiatric or somatic disease other than PD.
5. Abuse of alcohol or drugs according to Alcohol Use Disorders Identification Test (AUDIT), and/or clinical judgment.
6. Epilepsy.
7. Cerebral bleeding or history of cerebral bleeding.
8. Pregnancy or breastfeeding (will be asked).
9. Claustrophobia.
10. Smoking or using tobacco including snuff.
11. Dominant left-hand.
12. Inoperated apparatus (e.g., pacemaker).
13. Aneurysm clips in the head.
14. Shunts in the head.
15. Grenade-splinter or metal-splinter in the body (e.g.,eyes).
16. Metal or electrodes in the body (e.g., temp-catheter, aortastent, cochleaimplant).
17. Comprehensive tooth-implants or prothesis.
18. Operated in the head.
19. Operated in the heart.
20. Swallowed a video-capsule.
21. Any other reason the investigator feels the subject is not suitable for participation in the study.

Patients with IBS

Inclusion Criteria:

1. Fulfilling ROME IV criteria upon recruitment
2. Minimum 5 year of IBS symptoms
3. Males or females aged 18-85 years
4. Signed informed consent

Exclusion criteria:

1. Other confirmed GI diseases (such as inflammatory bowel diseases) or PD
2. Concurrent or recent treatment with antibiotics (< 12 weeks).
3. Concurrent or recent (< 4 weeks) use of nutritional supplements or herb products affecting intestinal function or mood (e.g. aloe vera, St. John´s Wort and probiotics/prebiotics).

3) Diagnosis of major psychiatric or somatic disease. 4) Abuse of alcohol or drugs according to Alcohol Use Disorders Identification Test (AUDIT), and/or clinical judgment.

5) Epilepsy. 6) Cerebral bleeding or history of cerebral bleeding. 7) Pregnancy or breastfeeding (will be asked). 8) Claustrophobia. 9) Smoking or using tobacco including snuff. 10) Dominant left-hand. 13) Inoperated apparatus (e.g., pacemaker). 14) Aneurysm clips in the head. 15) Shunts in the head. 16) Grenade-splinter or metal-splinter in the body (e.g.,eyes). 17) Metal or electrodes in the body (e.g., temp-catheter, aortastent, cochleaimplant).

18) Comprehensive tooth-implants or prothesis. 19) Operated in the head. 20) Operated in the heart. 21) Swallowed a video-capsule. 25) Any other reason the investigator feels the subject is not suitable for participation in the study.

Healthy controls:

Inclusions criteria:

1. Males or females aged 18-85
2. Signed informed consent

Exclusion criteria:

1. Concurrent or recent treatment with drugs affecting intestinal microbiota, function or mood, e.g., antidepressants (< 12 weeks), antibiotics (< 12 weeks)
2. No on going GI symptoms
3. Concurrent or recent (< 4 weeks) use of nutritional supplements or herb products affecting intestinal function or mood (e.g. aloe vera, St. John´s Wort and probiotics/prebiotics).
4. Diagnosis of major psychiatric or somatic disease.
5. Abuse of alcohol or drugs according to Alcohol Use Disorders Identification Test (AUDIT), and/or clinical judgment.
6. Recent (< 4 weeks) intake of proton pump inhibitors, PPI (e.g., omeprazol).
7. Epilepsy.
8. Cerebral bleeding or history of cerebral bleeding.
9. Pregnancy or breastfeeding (will be asked).
10. Claustrophobia.
11. Smoking or using tobacco including snuff.
12. Dominant left-hand.
13. Inoperated apparatus (e.g., pacemaker).
14. Aneurysm clips in the head.
15. Shunts in the head.
16. Grenade-splinter or metal-splinter in the body (e.g., eyes).
17. Metal or electrodes in the body (e.g., temp-catheter, aortastent, cochleaimplant).
18. Comprehensive tooth-implants or prothesis.
19. Operated in the head.
20. Operated in the heart.
21. Swallowed a video-capsule.
22. Regular intake of anti-inflammatory medication (including NSAIDs).
23. Any other reason the investigator feels the subject is not suitable for participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson patients will be recruited from the neurological department at Örebro University hospital by neurologist.
  Patients with IBS will be recruited from the gastroenterology deparments at Örebro University hospital by gastroenterologist.
  Healthy controls will be recruited via local advertisements or from previous study pools.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Presence of alpha-synuclein | Stored samples collected from a one day visit will be continously analysed during the 5 year project
  Alpha-synuclein is the hallmark protein of Parkinson's disease and the presence of this protein will be detected with immunoflourescence in colonic tissues

SECONDARY OUTCOMES:
Intestinal permeability | 1 day
  Colonic permeability measured by biopsies mounted in Ussing chambers
Mucosal ultrastructure: cell activation | Stored samples collected from a one day visit will be continously analysed during the 5 year project
  Morphologic quantification of cell size and granule density using Electron microscopy
Mucosal ultrastructure: cell-to-cell interaction | Stored samples collected from a one day visit will be continously analysed during the 5 year project
  Quantitative measurement of distance between cells to interpolate cell-to-cell interaction using Electron microscopy
Microbiota composition | Stored samples collected from a one day visit will be continously analysed during the 5 year project
  Analysis of faecal microbiota composition and function (metagenomics)
Metabolomics | Stored samples collected from a one day visit will be continously analysed during the 5 year project
  Metabolomic analysis of inflammatory markers, sex hormones and enviromental pollutants in blood and faeces
Brain function | 1day
  Structural and functional alterations in the brain and brainstem using functional magnetic resonance imaging
Aggregation potential of alpha-synuclein | Stored samples collected from a one day visit will be continously analysed during the 5 year project
  Measure the potential of alpha-synuclein to form aggregates in colonic biopsies
Platelet aggregation | 1 day
  Platelets will be isolated from blood samples and run on an aggregometer to elcuidate platelet aggregation potential
Immunophenotyping | 1 day
  Lamina propria lymphocytes will be characterised for their immune-neurophenotype using flow cytometry
Gastrointestinal Symptoms Rating Scale - Irritable Bowel Syndrome version (GSRS-IBS) | 1 day
  The Gastrointestinal Symptoms Rating Scale (GSRS) evaluates gastrointestinal (GI) symptoms based on the 5 domains diarrhoea, constipation, reflux, indigestion and abdominal pain. The symptoms are assessed with 15 items, ranging in scores 1 to 7 depending on their severity. A score of 1 represents "no problems" and score 7 represents "severe problems". The severity of symptoms may be defined as no problems (1 point), mild (1-2 points), moderate (2-4 points), and severe (4-7 points). The scores for each domain was calculated as the mean score of each corresponding item while the mean total GSRS score reflects the general severity of GI symptoms.
Irritable bowel syndrome- symptom severity scale (IBS-SSS) | 1 day
  This scale evaluates five aspects of IBS during a 10-day period: abdominal pain, distension, stool frequency and consistency and interference with daily life. Each item is scored on a visual analogue scale from 0 to 100 and the sum is the total score. The scale is responsive to treatment and has good validity.
Food Frequency Questionnaire (FFQ) | 1 day
  The dietary pattern will be assessed through a food frequency questionnaire that has been validated in a Swedish population. The questionnaire includes 174 foods and drinks and estimates the dietary pattern during one year. This is a common way to evaluate eating habits and in this way, evaluation of the microbiota composition in relation to dietary patterns is possible to assess.
Hospital Anxiety and Depression Scale (HAD) | 1 day
  The Hospital Anxiety and Depression Scale (HADS) was used to evaluate the psychological distress of study participants.This questionnaire consists of 14 items subdivided in two subscales for the assessment of anxiety or depression. The total score is used as a measure of general psychological distress. The minimum score is 0 and the maximum score is 21. A score > 8 on respective subscales indicates a significant level of anxiety or depression.
Perceived Stress Scale (PSS) | 1 day
  The perceived stress scale (PSS) consists of 10 items, including a number of direct questions about current levels of experienced stress. The respondent answers how often a certain emotion has been present during the past month. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Each item is rated on a 5-point scale ranging from never (0) to almost always (4). The questions in this scale ask about the responders feelings and thoughts during the last month. In each case the questionnaire requires the respondent to indicate by circling how often they felt or thought a certain way.
MDS Clinical Diagnostic Criteria for Parkinson's Disease | 1 day
  The MDS criteria use a two-step process of PD diagnosis. First, parkinsonism is defined (as bradykinesia in combination with either rest tremor, rigidity, or both). Once diagnosed, the criteria then define whether this parkinsonism is attributable to Parkinson's disease. Not scale-based.
Hoehn and Yahr scale/stages (Modified scale) | 1 day
  The Hoehn and Yahr scale is one of the most commonly and most widely used scale to describe severity in stages 1-5 of Parkinson's disease worldwide. The modified form includes 0.5 increments.
Clinical Impression of Severity Index for Parkinson's disease (CISI-PD) | 1 day
  The CISI-PD scale provides a clinical judgment on Parkinson's disease (PD) severity based on motor symptoms and complications, cognitive status, and disability. For each component, the score ranges from 0 (normal) to 6 (very severe). A brief definition is attached to each rank, and the sum of these four items yields a global index ranging from 0 to 24 points.
Non-Motor Symptoms Questionnaire | 1 day
  An instrument to assess wide range of non-motor symptoms based on list of 30 items by answering with: Yes, Don't know, No. This instrument does not provide an overall score of disability and is not a graded or rating instrument. Instead, it is a screening tool designed to draw attention to the presence of non-motor symptoms and initiate further investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, PhD/MD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Campus USÖ, Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No